CLINICAL TRIAL: NCT05792514
Title: The Reliable Nutritional Risk Screening Tools in Children Aged (2-5) Years Old Admitted to Assiut University Children Hospital
Brief Title: The Reliable Nutritional Risk Screening Tools
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Endy Mohammed Rashad, EMohammedRashad, Assiut University
Other Study IDs: malnutrition in children
Record Dates: First submitted 2023-02-26; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: stong,stamp,pyms — STRONG(screening tool for risk of nutritional status and growth) STAMP(screening tool assessment of malnutrition in pediatrics) PYMS
  Other Names: screening tools for malnutrition

SUMMARY:
* assess the subjective global validity and reliability of using The Pediatric Yorkhil Malnutrition Score (PYMs) and merits of using the Screening Tool for Risk on Nutritional status and Growth (STRONGkids) as a nutrition screening tool
* correlate it with the severity of their nutritional derangements in comparison to the Screening Tool for the Assessment of Malnutrition in Pediatrics (STAMP)in hospitalized Egyptian children aged (2-5)years in Assiut University Children Hospital (AUCH).

DETAILED DESCRIPTION:
Malnutrition is responsible for around 3.1 million child deaths annually in low and middle income countries,the malnutrition is involved in about 45% of under-five children deaths in numerous developing countries.

Malnutrition is associated with negative outcomes for inpatients, including increased risks of infections , increased muscle loss , impaired wound healing, longer hospital stay and increased morbidity and mortality .

Malnutrition may be responsible for delayed recovery and need for intensive nursing care, thus increasing the cost of hospitalization .

Nutritional support for inpatients has made progress and it is provided systematically through multidisciplinary nutritional support teams (NSTs) in most hospitals. The first step to run and manage the NST effectively and efficiently in each hospital may be proper screening and selection of the patients who are at risk of malnutrition requiring nutritional support during hospitalization Routine nutritional screening is rarely carried out in pediatric patients because of the lack of a simple and properly validated nutritional screening tool. The current practice of identifying children at risk of malnutrition is reliant on interpretation of anthropometric data and clinical judgement; the reliability of which is dependent on nutritional knowledge of pediatricians .

Severe cases of malnutrition are easily recognized; however, the identification of children with lesser degrees of malnutrition or at risk of malnutrition, which is also important, is not as easily achieved.

ELIGIBILITY:
Inclusion Criteria:

* all patients at the age of 2-5 years admitted in Assiut university children's hospital

Exclusion Criteria:

* no

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all patients at the age of 2-5 years admitted in Assiut university children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
the reliable nutritional risk screening tools in diseased children aged (2_5) years old admitted to Assiut University Children Hospital | 2 years
  asses the merits of using the Screening Tool for Risk on Nutritional status and Growth (STRONGkids) as a nutrition screening tool
the Screening Tool for the Assessment of Malnutrition in Pediatrics | 2 years
  asses the merits of using the the Screening Tool for the Assessment of Malnutrition in Pediatrics (STAMP) in hospitalized Egyptian children aged (2-5)years in Assiut University Children Hospital (AUCH).
using The Peduatric Yorkhil Malnutrition score | 2 years
  asses the subjective global validity and reliability of using The Pediatric Yorkhil Malnutrition Score (PYMs) in hospitalized Egyptian children aged (2-5)years in Assiut University Children Hospital (AUCH).

REFERENCES:
- See also: 1. ELSARY A.Y., ABD EL-MOKTADER A.M., ELGA MEEL A., MOHAMMED W.S., MASOUD M. and ABD EL-HALEEM N.G.: Nutritional survey among under five children at Tamyia district in Fayoum, Egypt. Int. J. Community Med. Public Health, 4 (6): 1813-8, 2017. Magnitude 2. — https://www.nature.com/articles/1602714